CLINICAL TRIAL: NCT04772053
Title: A Global, Molecular Disease Characterization Initiative (MDCI) in Oncology Clinical Trials
Brief Title: Molecular Disease Characterization Initiative (MDCI)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated for reasons pertaining to feasibility
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 213299
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer, Non-Small Cell; Neoplasms
Keywords: Tumor biopsy; Molecular Disease Characterization Initiative; Oncology; Clinical trial
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants undergoing tumor biopsy (Experimental)
  Interventions: Procedure: Tumor biopsy

INTERVENTIONS:
Procedure: Tumor biopsy — Archived or fresh tumor biopsy samples will be collected.

SUMMARY:
This is a single arm interventional molecular analysis study with no administration of investigational product and no masking. This multicenter study will involve participants with advanced/metastatic disease for the purpose of collecting tumor tissue and blood samples for broad molecular analysis and examining the expression of specific biomarkers using validated clinical assays.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a candidate for molecular screening for a GlaxoSmithKline (GSK) precision therapeutic clinical study (the Intended Treatment Protocol) that is being conducted in parallel at or nearby the MDCI recruitment site.
* Participant is willing to travel to a site recruiting for the intended GSK treatment protocol (or alternative treatment protocol), if feasible, and if, in the investigator's opinion, the participant would benefit from enrolment into the intended GSK treatment protocol at an alternative clinical site.
* Participants with confirmed advanced/metastatic diagnosis of solid malignancy in one of the following disease-areas: Non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), Breast, ovarian, and colorectal cancer (CRC).
* Participants with life expectancy of greater than (>) 6 months.
* Participants who are able to provide blood samples.
* Participants who are able to provide an archival formalin-fixed paraffin-embedded (FFPE) tumor specimen from a current lesion/most current setting (from no more than 2 years ago). If an archival tumor specimen is not available, surplus tissue from standard of care procedures is acceptable before fresh biopsy may be obtained.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP) or Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of less than [<]1 percent [%] per year), preferably with low user dependency; A WOCBP must have a negative highly sensitive pregnancy test (urine or serum) as required by local regulations) within 24 hours before tumor biopsy; and if a urine test cannot be confirmed as negative (for example, an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Participants capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).

Exclusion Criteria:

* Participants with Eastern Cooperative Oncology Group (ECOG) Performance Status >2.
* Participants with history of myocardial infarction, acute inflammatory heart disease, unstable angina, or uncontrolled arrhythmia within the past 6 months.
* For female participants, pregnancy.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with the participant's safety, obtaining informed consent or compliance to the screening study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Nashville, Tennessee, United States
- GSK Investigational Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated for reasons pertaining to feasibility.
Groups:
- Participants Who Underwent Tumor Biopsy: Participants with advanced/metastatic diagnosis of malignancy disease underwent tumor biopsy.
Period: Overall Study
Arm/Group | Participants Who Underwent Tumor Biopsy
Started | 6
Completed | 0
Not Completed | 6
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 3
Not completed — Study Terminated by Sponsor | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Who Underwent Tumor Biopsy
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 58.2 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Inducible T-cell Co-Stimulator (ICOS) Status
Description: Blood samples were collected for clinical biomarker testing and a tumor specimen was collected as per tumor specimen collection requirements. The specimen was evaluated by immunohistochemistry (IHC) to determine the expression of tumor specific antigens and immune markers. The ICOS is the biomarkers and data for participants with its positive status has been presented.
Time Frame: Up to approximately 17 months
Population: Enrolled population included all participants who signed the informed consent form (ICF) and met inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Underwent Tumor Biopsy
Number analyzed (Participants) | 6
Participants | 2

2. Primary Outcome: Number of Participants With Positive New York Esophageal Squamous Cell Carcinoma 1 (NY-ESO-1)/Cancer Testis Antigen 2 (LAGE-1a) Status
Description: Blood samples were collected for clinical biomarker testing and a tumor specimen was collected as per tumor specimen collection requirements. The specimen was evaluated by immunohistochemistry (IHC) to determine the expression of tumor specific antigens and immune markers. The NY-ESO-1 and LAGE-1a are biomarker and data for number of participants with its positive status has been presented.
Time Frame: Up to approximately 17 months
Population: Enrolled population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Underwent Tumor Biopsy
Number analyzed (Participants) | 6
Participants | 1

3. Primary Outcome: Number of Participants With Positive Programmed Death Protein 1 Ligand (PD-L1) Status
Description: Blood samples were collected for clinical biomarker testing and a tumor specimen was collected as per tumor specimen collection requirements. The specimen was evaluated by immunohistochemistry (IHC) to determine the expression of tumor specific antigens and immune markers. The PD-L1 is a biomarker and data for number of participants with its positive status has been presented.
Time Frame: Up to approximately 17 months
Population: Enrolled population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Who Underwent Tumor Biopsy
Number analyzed (Participants) | 6
Participants | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected maximum up to approximately 17 months.
Description: Enrolled population included all participants who signed the informed consent form (ICF) and met inclusion criteria
Arm/Group | Participants Who Underwent Tumor Biopsy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Underwent Tumor Biopsy (N=6)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Who Underwent Tumor Biopsy (N=6)
Asthenia (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT04772053/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT04772053/SAP_001.pdf